CLINICAL TRIAL: NCT02629211
Title: Initial Experience With a Novel Single-Balloon Enteroscopy System in Children With IBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Smart Medical Systems Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AB 17701
Record Dates: First submitted 2015-12-07; First posted 2015-12-14 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease
Keywords: Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Single-Balloon Enteroscopy; NaviAid AB™ Device; NaviAid AB™ Procedure; AB Device; Pediatric IBD; Pediatric Enteroscopy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NaviAid™ AB (Experimental): NaviAid™ AB device procedure
  Interventions: Device: NaviAid™ AB

INTERVENTIONS:
Device: NaviAid™ AB — NaviAid™ AB Procedure

SUMMARY:
To evaluate the safety and efficacy of the NaviAid™ AB in children with known or suspected IBD.

DETAILED DESCRIPTION:
In 15%-25% of diagnosed inflammatory bowel disease (IBD) cases, disease manifestation begins before the age of 18. IBD primary includes Crohn's disease (CD) and ulcerative colitis (UC). Studies have shown that the current incidence of pediatric IBD ranges from 4-7 cases per 100,000, worldwide. Early and accurate diagnosis of IBD is important for correct prognosis, course of disease, therapeutic decisions and follow-up. Complete diagnostic work-up is key to proper diagnosis in patients.Early diagnosis of IBD and differentiation between UC and CD can be difficult in children. The major issues that face pediatric IBD today include accurate disease classification, unknown extent of disease, complete bowel visualization, inability to reach depth of findings, and biopsy retrieval for diagnostic work-up.

The NaviAid™ AB device presents a new and unique concept that helps overcome these short comings of IBD diagnosis and treatment. Through repetitive inflation and deflation of the NaviAid™ AB, the endoscope can be swiftly advanced deep into the small bowel via the proximal or distal route, allowing for complete visualization of the small bowel and easy biopsy sampling for histopathology. As a result, subsequent diagnoses can influence proper action for further treatment and therapy for the patient. Although many studies have reported on the safety and efficacy of balloon enteroscopy in adults with IBD, further investigation of the value of balloon enteroscopy in pediatric patients with known or suspected IBD is still required.

This is a single-center, non-randomized open-label study intended to evaluate the safety and efficacy of the NaviAid™ AB device during small bowel enteroscopy in children with known or suspected IBD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages 8-18
2. Patients with known or suspected IBD (including Crohn's disease or ulcerative colitis).
3. The patient/parent of patient must understand and provide written consent for the procedure.

Exclusion Criteria:

1. Subjects with known coagulation disorder;
2. Subjects with known hernia;
3. Subjects with suspected stricture or stenosis;
4. Any patient condition deemed too risky for the study by the investigator
5. Subjects who are currently enrolled in another clinical investigation.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-01 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Number of serious adverse events | Subjects will be followed up with in 72 hours following the procedure.
  Patients will be followed up during the study period (3 hours) and once again 48-72 hours following the procedure. At both times, serious adverse events will be assessed.

SECONDARY OUTCOMES:
Number of findings | Up to 14 days (histology)
  Histology results will be used to assess this outcome
Procedural times | During procedure
Depth of insertion | During procedure
Ease of use | During procedure
  Ease of use will be scored using a scale of "Easy" Neutral" or "Difficult"
Classification of disease | Up to 14 days (histology)
  Histology results will be used to assess this outcome
Extension of disease | Up to 14 days (histology)
  Histology results will be used to assess this outcome

CONTACTS AND LOCATIONS:
Overall Officials: Efrat Broide, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Tzrifin, Israel

REFERENCES:
- [Derived] Broide E, Shalem T, Richter V, Matalon S, Shirin H. The Safety and Feasibility of a New Through-the-scope Balloon-assisted Enteroscopy in Children. J Pediatr Gastroenterol Nutr. 2020 Jul;71(1):e6-e11. doi: 10.1097/MPG.0000000000002706. PMID 32187142